CLINICAL TRIAL: NCT02156102
Title: Insights Into Microbiome and Environmental Contributions to Sickle Cell Disease and Leg Ulcers
Brief Title: Insights Into Microbiome and Environmental Contributions to Sickle Cell Disease and Leg Ulcers Study (INSIGHTS Study)
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140125; 14-HG-0125
Record Dates: First submitted 2014-06-04; First posted 2014-06-05 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-04

CONDITIONS: Genetic Disease; Genomics
Keywords: Genetic Disorders; Health contributors; Multifactorial; African American; African; Natural History
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Microbiome with active Leg Ulcer: We will recruit and obtain microbiome samples from male or female adult participants with active leg ulcers and sickle cell disease.
- Microbiome with no active Leg Ulcer: We will recruit and obtain microbiome samples from male or female adult participants without active leg ulcers but do have sickle cell disease.
- Non-microbiome participants: We will recruit but not obtain microbiome samples from participants with sickle cell disease

SUMMARY:
Background:

- People with sickle cell disease and other blood disorders sometimes get chronic leg ulcers. These are wounds that develop on the skin and don t go away. Current treatments do not work very well, so researchers want to learn more about why the ulcers happen. They want to find out which bacteria may cause it, and if external factors play a role.

Objective:

- To study social and environmental factors of sickle cell disease and the causes of sickle cell disease leg ulcers.

Eligibility:

- People age 18 and older who have sickle cell disease or another red cell disorder, with or without an active leg ulcer.

Design:

* Participants will have a medical history and clinical evaluation. They will also have blood drawn.
* Participants will complete questionnaires about their life, health, environment, stress, and other topics.
* Participants may provide a small sample of hair.
* Participants will be asked to collect a small amount of saliva.
* Participants with leg ulcers will have their skin microbiome sampled. The microbiome is all of the microbes (bacteria and and/or fungi) and their genes in and on the body. Researchers will use swabs to collect skin samples. Photographs will be taken of the skin sample area.
* Some participants without leg ulcers also will have their skin microbiome sampled.
* Some participants who have their skin microbiome sampled will return for a second visit. At this visit, their microbiome will be resampled. It will take place more than 30 days after the first visit.

DETAILED DESCRIPTION:
Study Description:

Leg ulcers are a serious and debilitating complication of sickle cell disease (SCD). This study will explore microbial, genomic, and environmental (social and physical) factors, that may influence the onset and progression of leg ulcer formation and delayed healing in individuals living with SCD. The etiology of SCD-associated leg ulcers is unclear, and we hypothesize that predisposition to developing leg ulcers is multifactorial. This multisite study is an exploratory study of the microbiome and environment of individuals living with sickle cell disease leg ulcers. The study s objective is to identify triggers that may be integral in leg ulcer onset and progression. The central goal of this study is to obtain an improved understanding of the participants clinical phenotype, leg ulcer microbiome and the psychosocial and environmental factors that may impact this complication.

Objectives:

Primary Objective:

Employ genomic approaches to characterize the skin microbiome in individuals living with SCD with and without leg ulcers.

Secondary Objective:

1. Employ social science research measures to identify psychosocial and physical environmental factors that impact quality of life in individuals living with SCD with and without leg ulcers.
2. Develop new measure of severity for SCD that integrates clinical outcomes and the quality of life of the participant.
3. Develop guidelines for researchers to address the needs of diverse and under-resourced groups in genetic research.

Endpoints:

Primary Endpoint:

To characterize the microbiome of leg ulcers in SCD.

Secondary Endpoints:

1. To characterize the phenotypic variation in SCD.
2. To identify similarities and differences of the microbial signatures of chronic diabetic foot ulcers and SCD leg ulcers.
3. To investigate physical and psychosocial environmental indicators that impact quality of life in individuals living with SCD with and without leg ulcers.
4. To determine if an association exists between the microbiome (microbial diversity) of SCD leg ulcers and the quality of life (psychosocial and physical environment) indicators of individuals with SCD leg ulcers.
5. To determine if an association exists between the microbiome (microbial diversity) of SCD leg ulcers and clinical phenotype of individuals with SCD leg ulcers.
6. To determine how leg ulcers influence one s physical function and one s perceptions of stigma and self-esteem.
7. To identify factors that are indicators of both quality of life and clinical severity of the participant.
8. To identify specific psychosocial and environmental factors related to resilience in our study population.
9. To investigate current practices and policies around the return of secondary findings in genome sequencing studies in under-resourced study participant populations, and to explore ethical and clinical policies for returning secondary findings by examining various practices within the research community.
10. To investigate SCD variation in phenotype, microbiome, physical and psychosocial environments in a cohort in Sierra Leone.
11. To compare similarities and differences in phenotype, microbiome, physical and psychosocial environments between U.S. and Sierra Leone cohorts.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will enroll up to four-hundred and fifty (N=450) participants in the microbiome sampling cohort. In addition to the 300 SCD leg ulcer microbiome participants, we will recruit up to an additional 200-250 SCD participants that will complete the clinical evaluation, (including blood sample) and survey instruments for a total of up to 550 participants at three sites, NIH (n=200) and MMC (n=100), and Sierra Leone (n=250).

Of the total participants, we will resample the microbiome of up to 75 individuals from each of the 3 initial sampling groups: SCD with, without and never had SCD leg ulcers. Of those 75 individuals who are sampled longitudinally, those with clinically interesting cases may be sampled at multiple intervals.

All sampling, surveys, and processing of samples will take place at the NIH Clinical Center the second site, MMC, or in Sierra Leone. All samples will be stored at NIH.

To be eligible to participate in this study, an individual must meet all of the following criteria:

* All subjects must have a diagnosis of sickle cell disease (HbSS, HgSC, HbSB 0 or HBSB+)
* Be at least 18 years old.
* Provide written informed consent.
* For the Qualitative phase: must have a recurrent, active, or single-occurrence presentation of a leg ulcer(s).
* For the resilience study analysis: cohort will be determined by the research team based on the results of part I of this analysis. For part I, the inclusion criteria are that the individual must have enrolled and completed the INSIGHTS study.

EXCLUSION CRITERIA:

Any individual that meets any of the following criteria during baseline evaluation will be excluded from the study:

* Pediatric population (<18 years old)
* Participants for microbiome study (only) who have received oral and/or topical antibiotics or antifungals < 2 weeks prior to enrolling in the study for leg ulcers (for those with leg ulcers only)
* Subjects presenting with clinically diagnosed bacterial infection (i.e. clinical appearance, clinical judgment, fever, redness around ulcer, purulent drainage etc.) at the site of ulceration. (This can only be diagnosed clinically by the research nurse during sampling

and is only applicable to those with leg ulcers only).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a descriptive study of individuals living with sickle cell diseases (SCD) with and without leg ulcers (accrual goal 550 participants). Leg ulcers are not observed in all individuals with SCD and we are interested in understanding why certain individuals develop leg ulcers. We will seek to include age-matched patients without leg ulcers for the microbiome phase of the study. We will recruit and sample male or female adult participants with ulcers, currently without leg ulcers, and those with no previous history of leg ulcers. To ensure we recruit an adequate number of participants with and without leg ulcers, we will rely on multiple recruiting methods, which will include posting flyers, social media advertisements, and/or referrals.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
The skin microbiome | Assessment occurs on date of visit.
  Employ genomic approaches to characterize the skin microbiome in individuals living with SCD with and without leg ulcers
The factors that impact quality of life | Assessment occurs on date of visit.
  Employ social science research measures to identify psychosocial and physical environmental factors that impact quality of life in individuals living with SCD with and without leg ulcers
Sickle Cell disease severity measure | Assessment occurs on date of visit.
  Develop new measure of severity for SCD that integrates clinical outcomes and the quality of life of the participant

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Koehly, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (3):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York
- University of Sierra Leone, College of Medicine and Allied Health Services, Freetown, Sierra Leone

REFERENCES:
- [Background] Minniti CP, Eckman J, Sebastiani P, Steinberg MH, Ballas SK. Leg ulcers in sickle cell disease. Am J Hematol. 2010 Oct;85(10):831-3. doi: 10.1002/ajh.21838. PMID 20872960
- [Background] Umeh NI, Ajegba B, Buscetta AJ, Abdallah KE, Minniti CP, Bonham VL. The psychosocial impact of leg ulcers in patients with sickle cell disease: I don't want them to know my little secret. PLoS One. 2017 Oct 18;12(10):e0186270. doi: 10.1371/journal.pone.0186270. eCollection 2017. PMID 29045487
- [Background] Crouch EM, Bonham VL, Abdallah K, Buscetta A, Vinces G, Heo M, Minniti CP. Nutritional supplement profile of adults with sickle cell disease. Am J Hematol. 2018 May 4:10.1002/ajh.25129. doi: 10.1002/ajh.25129. Online ahead of print. No abstract available. PMID 29726579
- [Derived] Abdallah KE, Cooper KE, Buscetta AJ, Ramirez HC, Neighbors HW, Bonham VL. An Examination of John Henryism in Adults Living with Sickle Cell Disease. J Racial Ethn Health Disparities. 2025 Aug;12(4):2335-2344. doi: 10.1007/s40615-024-02054-5. Epub 2024 Jul 8. PMID 38977655
- [Derived] Raymond MB, Cooper KE, Parker LS, Bonham VL. Practices and Attitudes toward Returning Genomic Research Results to Low-Resource Research Participants. Public Health Genomics. 2021;24(5-6):241-252. doi: 10.1159/000516782. Epub 2021 Jul 6. PMID 34229325
- [Derived] Desine S, Eskin L, Bonham VL, Koehly LM. Social support networks of adults with sickle cell disease. J Genet Couns. 2021 Oct;30(5):1418-1427. doi: 10.1002/jgc4.1410. Epub 2021 Apr 12. PMID 33847032
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-HG-0125.html